CLINICAL TRIAL: NCT06745479
Title: Promoting Adaptive Decision-Making in Schizophrenia Through Improved Evidence Integration: A Combined Neuroimaging and Experience Sampling Study
Brief Title: Decision-Making in Schizophrenia: A Combined Neuroimaging and Experience Sampling Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Harold Zald, Ph.D., Henry Rutgers Term Professor of Psychiatry, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2023001193; R21MH135329-01A1 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Control Subjects
Keywords: Cognitive Strategy; Emotion Regulation; Psychosis; Schizophrenia; functional MRI
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): There is only 1 arm in this study. In this arm of the study, participants are instructed to implement a cognitive strategy (i.e., way of thinking) during 1/2 of the trials of a behavioral, gambling task. On the other 1/2 of the trials they behave naturally without implementing the cognitive strategy.
  Interventions: Behavioral: Positive Emotion Upregulation

INTERVENTIONS:
Behavioral: Positive Emotion Upregulation — Participants will identify personal goals or activities that they would like to engage in more and describe these goals/activities in a written format with research staff. Participants will then complete a gambling task during functional MRI scanning. Prior to making some gambling decisions, participants are instructed to mentally imagine achieving a goal or engaging in an enjoyable activity. Prior to the other decisions participants are instructed to respond naturally (i.e., not use the cognitive strategy).

SUMMARY:
The goal of this clinical trial is to learn if attention and ways of thinking impact decision-making and brain processes related to decision-making in people with schizophrenia or schizoaffective disorder relative to people without either condition. It will also learn how brain functioning during decision-making relates to real-world decisions made during daily life. The main questions it aims to answer are:

* Does paying attention to specific information impact decision-making and brain processes?
* Does thinking in a certain way according to specific 'thinking strategies' improve brain processes related to decision-making?
* Does brain functioning during decision-making relate to real-world choices to engage in activities?

Researchers will compare brain functioning and decision-making on computer tasks of gambling after participants have been trained to use a positive thinking strategy. They will compare what is different in the brain and behavior when participants use this strategy and when they do not. Participants will also answer brief surveys about activities and feelings for a week in their daily lives.

Participants will:

* Complete several hours of clinical interviewing, cognitive tests, and surveys of about symptoms, experiences, and personality
* Complete computer tasks about gambling decisions during MRI brain scanning and while having their visual attention measured using eye-tracking
* Complete brief surveys about their activities and feelings 5 times a day for 1 week using a cell phone. Each survey only take several minutes.

DETAILED DESCRIPTION:
This study aims to identify how attention and different ways of thinking impact decision making and brain activity. We are specifically examining how these factors differ between individuals with schizophrenia or schizoaffective disorder and individuals who do not have these conditions. We are also investigating how brain functioning during decision-making tasks correlates with real-world decisions recorded in everyday life. This ongoing study utilizes functional MRI brain imaging, eye-tracking, and daily event-sampling self-reports to identify whether there are differences in decision-making tendencies between groups of participants.

ELIGIBILITY:
Inclusion Criteria

The following criteria apply to all subjects:

1. Between ages of 18-45.
2. Have capacity to provide informed consent
3. Fluent communication in English
4. Willingness and ability to follow study requirements, as evidenced by an ability to provide written or virtual informed consent and read, and complete, study procedures.
5. Cognitive ability to understand tasks and estimated IQ greater than 70.

The following criteria apply to subjects with schizophrenia:

1. Primary diagnosis of schizophrenia or schizoaffective disorder

The following additional criteria apply to subjects without schizophrenia:

1. Inclusion based on subject matched to psychiatric group based on age, sex, race/ethnicity, and education level.

Exclusion Criteria

The following criteria apply to all subjects:

1. Self-disclosed or noticeable intoxication from alcohol or illicit drugs (e.g., arriving to participate in the study drunk/high)
2. Self-disclosure of consistent current substance use other than nicotine, alcohol, or cannabis (e.g. cocaine, heroin).
3. Many-year history of severely disordered substance use other than nicotine/tobacco (determined via interview)
4. Significant physical health disorder, robust physical health conditions, neurological disease/disorder (e.g., Parkinson's, history of strokes).
5. History of traumatic brain injury, head injury resulting in loss of consciousness for an extended duration or with noted neurobehavioral consequences.
6. Electroconvulsive therapy within one month of participation.
7. History of seizures or epilepsy.
8. Currently untreated or unstable psychiatric and medical conditions.
9. Intellectual disability
10. Contra indications for MR imaging (detailed below)

The following additional criteria apply to subjects without schizophrenia:

1. Pervasive history of problematic substance use (other than nicotine or alcohol) as defined by meeting DSM-5 criteria for a substance use disorder.
2. Diagnosis of, or first-degree relative with, significant psychiatric disorder (e.g., bipolar disorder, psychotic disorder, or Cluster A personality disorder).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Nucleus Accumbens Brain Activation | Single timeframe during 1.5 hours of MRI scanning and behavioral task completion.
  Brain activation in the nucleus accumbens (ventral striatum) measured via functional magnetic resonance imaging (fMRI) on trials that are preceded by the cognitive regulation strategy relative to trials without the cognitive regulation strategy.
Gambling Choice Behavior | Single timeframe during 1.5 hours of MRI scanning and behavioral task completion.
  Risky reward pursuit, defined as gamble choices on trials that are preceded by the cognitive regulation strategy relative to trials without the cognitive regulation strategy.

SECONDARY OUTCOMES:
Brain Activation and Functional Connectivity | Single timeframe during 1.5 hours of MRI scanning and behavioral task completion
  Brain activation and functional connectivity in areas across the whole brain measured via functional magnetic resonance imaging (fMRI) on trials that are preceded by the cognitive regulation strategy relative to trials without the cognitive regulation strategy.

CONTACTS AND LOCATIONS:
Overall Officials: David Zald, PhD, Principal Investigator — Rutgers University
Locations (1):
- Center for Advanced Human Brain Imaging Research, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Unless consent is withdrawn by participants at the individual level, data will be uploaded to the National Data Archive (NDA) in accordance with their timelines, data cataloguing criteria, and rules for data access requests.
Time Frame: Data will be uploaded in accordance with National Data Archive (NDA) data upload timelines and procedures.
Access Criteria: Data will be accessible via the National Data Archive (NDA) according to established data request procedures.
URL: https://nda.nih.gov/